CLINICAL TRIAL: NCT01075594
Title: Centralized Pan-Bulgarian Survey on the Undertreatment of Hypercholesterolemia
Brief Title: Study of Undertreatment of Patients With Dyslipidemia in Bulgaria
Acronym: CEPHEUS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Other Study IDs: NIS-CBG-CRE-2009/1
Record Dates: First submitted 2010-02-19; First posted 2010-02-25 (Estimated); Last update posted 2010-09-10 (Estimated); Status verified 2010-09

CONDITIONS: Dyslipidemia
Keywords: Dyslipidemia; Target cholesterol; Undertreatment
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: None Retained — whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with dyslipidemia on lipid lowering therapy

SUMMARY:
The purpose of this study is to establish the proportion of Bulgarian patients on lipid-lowering pharmacological treatment reaching the LDL-C goals according to the Fourth Joint European Task Force guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Lipid lowering drug treatment for at least 3 months, with no dose change for a minimum of 6 weeks
* Signed Informed Consent

Exclusion Criteria:

* Informed Consent not provided

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2010-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The number and percentage of patients achieving the LDL-C goals, according to the Fourth Joint European Task Force guidelines | 6 months - one visit only, no follow-up visits

SECONDARY OUTCOMES:
The number and percentage of subjects achieving the LDL-C goals, according to the Fourth Joint European Task Force guidelines for several subject subsets | 6 months - one visit only, no follow-up visits
The number and percentage of subjects achieving LDL-C goals according to the NCEP ATP III / 2004 updated 2004 NCEP ATP III guidelines, overall and for several subject subsets | 6 months - one visit only, no follow-up visits
The number and percentage of subjects achieving the non HDL-C goals according to the NCEP ATP III/updated 2004 NCEP ATP III/national guidelines [<130mg/dL (3,37mmol/L)], in the following sub-population: patients with fasting triglycerides >200 mg/dL | 6 months - one visit only, no follow-up visits

CONTACTS AND LOCATIONS:
Locations (15):
- Bulgaria (15):
  - Research Site, Blagoevgrad
  - Research Site, Burgas
  - Research Site, Haskovo
  - Research Site, Montana
  - Research Site, Pazardzhik
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Shumen
  - Research Site, Sliven
  - Research Site, Smolyan
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
  - Research Site, Veliko Tarnovo